CLINICAL TRIAL: NCT01095861
Title: Comparison of Parker Flex-Tip Endotracheal Tube to Standard Endotracheal Tube: A Randomized Controlled Trial
Brief Title: Comparison of Parker Flex-Tip Endotracheal Tube to Standard Endotracheal Tube
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Timothy P Turkstra, University of Western Ontario
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R-09-126; 16016 (Other: REB)
Record Dates: First submitted 2009-09-02; First posted 2010-03-30 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2011-08

CONDITIONS: Endotracheal Intubation
Keywords: endotracheal tube

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FlexTip ETT (Experimental): FlexTip ETT
  Interventions: Device: FlexTip ETT (Parker FlexTip/GlideScope FlexTip)
- Control (Placebo Comparator): Standard Flexible ETT Mallinckrodt Hi-Lo cuffed tracheal tube Catalog # 86114 Mallinckrodt, ST. Louis, MO, 63134
  Interventions: Device: Control - standard flexible ETT (Mallinckrodt)

INTERVENTIONS:
Device: FlexTip ETT (Parker FlexTip/GlideScope FlexTip) — FlexTip ETT used for endotracheal intubation
  Other Names: Parker FlexTip; GlideScope FlexTip
  Arms: FlexTip ETT
Device: Control - standard flexible ETT (Mallinckrodt) — Control - standard flexible ETT
  Mallinckrodt Hi-Lo cuffed tracheal tube, Catalog # 86114, Mallinckrodt, ST. Louis, MO, 63134
  Arms: Control

SUMMARY:
Patients presenting for elective surgery requiring tracheal intubation will be randomized to one of two different endotracheal tubes (ETT).

DETAILED DESCRIPTION:
The post-operative complication of a sore throat after endotracheal intubation is unfortunately common, with estimates ranging from 15-50%. Most estimates are in the order of 35-45%.(McHardy 1999, Higgins 2002) There is evidence that many patients do not report sore throat and/or vocal changes unless directly asked because surgical pain is more prominent and many patients may be unaware that intubation completed as part of the general anesthetic. (Harding 1987)

The Parker FlexTip® endotracheal tube (ETT) is formulated with a softer plastic at the distal tip as well as a laterally curved profile to reduce trauma during ETT advancement. (Makino 2003) This ETT has been shown to be faster during fibreoptic intubation, but complication of sore throat was not examined. (Kristensen 2003)

Our previous study (Jones 2007) demonstrated that modification of anesthetic techniques could reduce the incidence of post-operative sore throat in patients undergoing naso-tracheal intubation. We will now study the Parker Flex-Tip ETT to see if its use can also reduce the incidence of sore throat in patients undergoing oro-tracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient scheduled for elective surgery.
* ETT is indicated for the procedure in the opinion of the attending anesthesiologist.

Exclusion Criteria:

* Any patients with known or probable difficult airways.
* Any patient requiring rapid sequence induction.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Sore throat | 48-72 hours
  Patients fill in a questionaire 48-72 hours after Surgery by a blinded data assessor.
  They are asked if they had a sore throat after their surgery. If so, they are asked to grade the sore throat as mild, moderate, or severe, when it was at its worst.
  Note: There is only one questionaire for both outcomes.

SECONDARY OUTCOMES:
Vocal changes | 48-72 hours
  Patients fill in a questionaire 48-72 hours after Surgery by a blinded data assessor.
  They are asked if they had vocal changes after their surgery. If so, they are asked to grade the vocal changes as mild, moderate, or severe, when the changes were at its worst. Patients are asked for one word to best characterise the vocal changes.
  Note: There is only one questionaire for both outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy P Turkstra, MD, M. Eng, Principal Investigator — Western University, Canada; Philip M Jones, MD, Principal Investigator — Western University, Canada
Locations (1):
- University of Western Ontario, London, Ontario, Canada

REFERENCES:
- [Derived] Turkstra TP, Smitheram AK, Alabdulhadi O, Youssef H, Jones PM. The Flex-Tip tracheal tube does not reduce the incidence of postoperative sore throat: a randomized controlled trial. Can J Anaesth. 2011 Dec;58(12):1090-6. doi: 10.1007/s12630-011-9592-5. Epub 2011 Nov 5. PMID 22057874